CLINICAL TRIAL: NCT06972147
Title: Prevalence and Description of FIRE (Food Induced Immediate Response of the Esophagus) in the Pediatric Population With Eosinophilic Esophagitis
Acronym: FIREO
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Other Study IDs: 49RC25_0086; CHU Angers (Other: CHU Angers)
Record Dates: First submitted 2025-03-14; First posted 2025-05-14 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-10

CONDITIONS: Eosinophilic Esophagitis
MeSH Terms: conditions — Eosinophilic Esophagitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- eosinophilic esophagitis: questionnary

SUMMARY:
A new clinical entity of eosinophilic esophagitis, Food Induced Immediate Response of the Esophagus or FIRE, has been described since 2020. Diagnostic criteria are not clearly established. Specific questioning is necessary for differential diagnosis, such as the oro-pharyngeal syndrome notably described in pollinics, or a mechanical blockage strictly speaking linked to esophagitis. The aim is to obtain epidemiological data on this entity.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 6 and under 18 years of age at the time of inclusion
* Follow-up in the allergology unit of Angers University Hospital for eosinophilic esophagitis

Exclusion Criteria:

* Patients or legal representative with severe communication or language comprehension difficulties
* Patients or legal representatives objecting to study participation

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patient follow-up in the allergology unit of Angers University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
diagnosis of FIRE syndrome | day 1
  symptoms such as pain, pressure, choking or narrowing, in the oesophagus or retrosternum, within 10 minutes of ingestion, lasting a maximum of 120 minutes, when a specific food is ingested

CONTACTS AND LOCATIONS:
Overall Officials: Anne HOPPE, Principal Investigator — University Hospital of Angers
Locations (2):
- France (2):
  - HOPPE Anne, Angers
  - CHU Lille, Lille

IPD SHARING:
Plan to Share IPD: Undecided